CLINICAL TRIAL: NCT01784354
Title: Acupressure in Raynaud's Phenomenon- A Pilot Study.
Brief Title: Acupressure for the Treatment of Raynaud's Phenomenon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Heather Gladue, DO, Principle Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00062868
Record Dates: First submitted 2013-01-18; First posted 2013-02-05 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Primary Raynaud's Phenomeon
MeSH Terms: interventions — Acupressure; Educational Status

ARMS (3):
- Education (Placebo Comparator): target education toward Raynaud's
  Interventions: Behavioral: education
- Acupressure (Active Comparator): acupressure- dilatation
  Interventions: Other: Acupressure dilatation
- Acupressure relaxation (Active Comparator): acupressure relaxation protocol
  Interventions: Other: Acupressure

INTERVENTIONS:
Other: Acupressure
  Arms: Acupressure relaxation
Other: Acupressure dilatation
  Arms: Acupressure
Behavioral: education
  Arms: Education

SUMMARY:
The use of acupressure will be compared to targeted Raynaud's education and will evaluate the' frequency, duration and pain of Raynaud's attacks.

DETAILED DESCRIPTION:
Using a Raynaud's condition score, severity of tingling, numbness and pain of attacks, the number of attacks and patient and physician visual analog scale we will assess the effect of acupressure.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Have Raynauds phenomenon, with at least 4 attacks in the last week
* on stable medications
* Willing to attend study visits

Exclusion Criteria:

* smoker
* have a history of stroke, heart attack or irregular heart rhythm
* uncontrolled blood pressure
* physical or mental illness that would interfere with participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Decrease in number of Raynaud's attacks | 1-2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States